CLINICAL TRIAL: NCT05685186
Title: A Longitudinal, Observational Study of Primary Ciliary Dyskinesia in Adults
Status: Active, not recruiting | Type: Observational
Sponsor: ReCode Therapeutics (Industry)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: RCTAX001
Record Dates: First submitted 2022-12-19; First posted 2023-01-13 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: PCD; Primary Ciliary Dyskinesia; Kartagener Syndrome
MeSH Terms: conditions — Ciliary Motility Disorders; Kartagener Syndrome | interventions — Spirometry; Mucociliary Clearance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PCD Cohort: The PCD cohort will include individuals who have a genetically confirmed diagnosis of PCD with 2 identified pathogenetic variants within 1 of 4 genetic/ultrastructural variants:
  * DNAI1 ODA defect
  * Other ODA defect
  * IDA-MTD defect, CCDC39 or CCDC40
  * Radial Spoke defect
  Interventions: Diagnostic Test: Spirometry; Diagnostic Test: Multiple Breath Washout (MBW); Diagnostic Test: Mucociliary Clearance (MCC); Diagnostic Test: CT of the chest; Diagnostic Test: MRI of the chest
- Healthy Volunteer Cohort: The healthy volunteer cohort will include health individuals.
  Interventions: Diagnostic Test: Spirometry; Diagnostic Test: Mucociliary Clearance (MCC); Diagnostic Test: MRI of the chest

INTERVENTIONS:
Diagnostic Test: Spirometry — To assess lung function
Diagnostic Test: Multiple Breath Washout (MBW) — To measure Lung Clearance Index (LCI)
  Groups: PCD Cohort
Diagnostic Test: Mucociliary Clearance (MCC) — To measure lung clearance after the inhalation of radiolabeled particles
Diagnostic Test: CT of the chest — Low radiation to assess structural lung disease
  Groups: PCD Cohort
Diagnostic Test: MRI of the chest — To assess lung function and structural lung disease

SUMMARY:
The goal of this observational study is to characterize clinical measures and biomarkers of airway disease in adults with primary ciliary dyskinesia (PCD) and in a group of healthy volunteers (HV) to establish normative values. Lung function, mucociliary clearance, radiological findings, and clinical findings will be assessed. Furthermore, quality of life will be assessed using QOL-PCD, a disease specific questionnaire.

DETAILED DESCRIPTION:
Primary ciliary dyskinesia (PCD) is a rare, genetically heterogeneous disease characterized by progressive upper and lower respiratory tract infections and inflammation caused by impaired mucociliary clearance (MCC). While longitudinal studies of children and adolescents with PCD have informed the early natural history of lung disease, there remains a knowledge gap in disease characteristics and progression in adults. There are no prospective published data evaluating the natural history of airway morbidity and mortality in adults, and little is known about the optimal clinical measures and biomarkers to evaluate disease progression. Cohort studies are needed to understand clinical measures and biomarkers across the lifespan of people with PCD, distinguish disease subtypes, and define endpoint variability. Natural history studies are critical for designing future clinical trials. New therapies have lagged in part due to lack of clear clinical biomarkers for adults.

The overarching goal is to characterize clinical measures and biomarkers of airway disease in adults with PCD. In addition, a subset of these clinical measures and biomarkers will be collected in a group of healthy volunteers (HV) to establish normative values.

ELIGIBILITY:
Inclusion Criteria:

* PCD diagnosis with confirmation of 2 identified pathogenic genetic variants within 1 of the following ultrastructure variants:
* DNAI1 ODA defect
* Other ODA defect
* IDA - MTD defect
* RS defect
* Informed consent

Exclusion Criteria:

* Are a current smoker (e-cigarette, tobacco, or marijuana)
* Are a former smoker who discontinued smoking <1 year prior to enrollment or has a cumulative 1+ pack-year smoking history
* Have a recent stable forced expiratory volume in one second (FEV1) <35% predicted
* Have contraindications for MRI studies (implanted devices/materials; inability to tolerate; claustrophobia or severe anxiety that would preclude MRI/imaging)
* Have had a significant clinical radiation exposure (as determined by the investigator) within the past 6 months. Potential participants who have had a chest CT within the past 6 months may be eligible to be enrolled and their clinical CT will be utilized as the baseline for this study
* Are pregnant or breastfeeding
* Have any comorbidities likely to impact lung function (e.g., complex congenital heart disease, severe scoliosis, diseases involving immune dysregulation, lung transplantation, lung lobectomy, end-stage renal disease, or poor overall health status).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals with a diagnosis of Primary Ciliary Dyskinesia and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-04-28 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Descriptive Analysis | From Baseline Through Week 52
  Descriptive statistical methods will be applied to analyze: lung function, measure % predicated (pp) FEV1. Absolute Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) Through Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Priya Ryali, Study Director — ReCode Therapeutics; Stephanie Davis, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States